CLINICAL TRIAL: NCT07146334
Title: Low Powered Colorectal Anastomosis After Rectal Excision : An Exploratory, Observational, Prospective, IDEAL Stage 2b International Cohort Study (OASIS)
Brief Title: Low Powered Colorectal Anastomosis After Rectal Excision (OASIS)
Acronym: OASIS
Status: Not yet recruiting | Type: Observational
Sponsor: Bordeaux Colorectal Institute (Other)
Responsible Party: Sponsor
Other Study IDs: B.C.I. 2025/01
Record Dates: First submitted 2025-07-31; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-07

CONDITIONS: Rectal Cancer; Surgery Indication
Keywords: rectal cancer; Transanal Transection and Single Staple anastomosis (TTSS); Double-stapled anastomotic (DS); mechanical anastomosis; rectal surgery; anastomotic leakage
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rectal surgery with powered mechanical anastomosis performed with DS or TTSS techniques: This is an international cohort (France and other international centers) which consists of including patients undergoing rectal surgery with powered mechanical anastomosis performed with DS or TTSS techniques.
  Surgeons at each center perform one or both techniques. When both types of stapling are possible, the choice of technique is made by the surgeon during the preoperative consultation, in the best interest of the patients, after a case-by-case assessment.

SUMMARY:
The objectiive of this prospective, international cohort is to compare two anastomotic techniques (DS vs TTSS) by collecting data during the surgery, and postoperatively (morbidity and functional outcomes).

The choice of technique is left to the discretion of the surgeon based on her/his practices.

DETAILED DESCRIPTION:
There are a variety of available anastomotic techniques to facilitate restorative surgery following total mesorectal excision (TME) for rectal cancer. However, there is no good quality evidence demonstrating the superiority of any single technique with regards to the potential sequalae of restorative surgery including anastomotic leakage and functional impact. Double-stapled anastomotic technique (DST) for colorectal anastomosis is the most widely used technique worldwide. An alternative to DST is the hand-sewn coloanal anastomotic (CAA) technique, which is traditionally reserved for patients with ultralow rectal tumours requesting restorative surgery or in cases of technical difficulties whereby a low colorectal anastomosis is converted to a coloanal anastomosis. More recently, the Transanal Transection and Single Staple anastomosis (TTSS) technique has been described. The TTSS technique has the potential to mitigate the difficulties encountered with DST and the potential complications and long-term functional sequalae encountered with handsewn anastomosis. Moreover, powered mechanical circumferential staplers represent a significant advancement in colorectal surgery, particularly in performing anastomosis following rectal excision. These devices are designed to provide consistent staple formation and controlled tissue compression, reducing the variability associated with manual stapling.

AL has a significant impact on clinical, patient-reported, and oncological outcomes. To mitigate the impact of AL a diverting stoma is routinely used to protect the distal anastomosis and facilitate anastomotic healing, with these stomas reversed once the integrity and patency of the distal anastomosis is confirmed. However, there is a significant complication profile associated with the routine use of diverting stomas. Through the incorporation of appropriate pre-operative risk stratification and careful post-operative surveillance a selective stoma strategy is associated with good clinical and functional outcomes.

The use of Double-stapled anastomotic technique (DST) or Transanal Transection Single-Stappled (TTSS) by laparoscopic or robotic approach, using or not a defunctionning stoma could not be separately tested in randomized trial.

In this exploratory, observational, prospective, IDEAL stage 2b International cohort study, we aim to include 400 patients with resection rectal and low powered colorectal anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patients with rectal cancer lower than 12 cm from the anal verge requiring either a stapling anastomosis below 7 cm from the anal verge,
* Patients with powered mechanical anastomosis (INTOCARE devices)
* Patients with no metastasis
* Patients operated on by mini-invasive rectal excision (laparoscopic, robotic or TaTME);
* Patients with or without defunctioning ileostomy;
* Patients with or without neoadjuvant treatment;
* Patient who benefits by medicare system;
* Signed and dated informed consent

Exclusion Criteria:

* Patients with handsewn anastomosis
* Patients with perforated rectal cancer or preoperative pelvic sepsis ;
* Patients with inflammatory bowel disease;
* Patients operated on in emergency ;
* Patients with extended-TME or pelvic exenteration;
* Pregnancy or breast feeding period
* Legal incapacity or physical, psychological social or geographical status interfering with the patient's ability to agree to participate in the study
* Persons deprived of liberty or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this exploratory, observational, prospective, IDEAL stage 2b International cohort study, we aim to include 400 patients with resection rectal and low powered colorectal anastomosis. This study is to compare two anastomotic techniques (DS vs TTSS) by collecting data during the surgery, and postoperatively (morbidity and functional outcomes).
  Surgeons at each center perform one or both techniques. When both types of stapling are possible, the choice of technique is made by the surgeon during the preoperative consultation, in the best interest of the patients, after a case-by-case assessment.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
To assess and compare the rate of anastomotic leakage at 1 month after rectal excision between double and single-stapling low colorectal anastomosis using advanced powered stapler | From the surgery to one month
  Proportion of anastomotic leakage (clinical and radiological) at 1 month after rectal surgery between double- and single-stapling low colorectal anastomosis using advanced powered stapler.

SECONDARY OUTCOMES:
Overall morbidity and mortality rates at 1 month | At 1 month after the end of the surgery
  Postoperative morbidity and mortality according Clavien-Dindo classification at 1 month
The rate of anastomotic leakage at 6 and 12 months after rectal surgery; | At 12 month after the end of the surgery
  Rate of defunctioning stoma at 1, 6 and 12 months after surgery;
Quality of life with QLQ C30 questionnaire | At 1, 6 and 12 months after rectal surgery
  The EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients.
  This is a patients self-rating questionnaire that measures five functional scales (physical, role, social, emotional, and cognitive) three symptom scales (fatigue, pain, nausea and vomiting) A global health status / QoL scale, and a number of single items assessing additional symptoms commonly reported by cancer patients (dyspnea, loss of appetite, insomnia, constipation and diarrhea) and perceived financial impact of the disease. Scores can be linearly transformed to provide a score from 0 to 100 REF. Higher scores represent better functioning on the functional scales and a higher level of symptoms of the symptom scales.
  9 dimensions will be assessed with: PF : Physical Functioning RF : Role Functioning CF : Cognitive Functioning EF : Emotional Functioning SF: Social Functioning FA : Fatigue PA : Pain NV : Nausea and Vomiting QL : Global health status
Quality of life with QLQ CR29 questionnaire | At 1,6 and 12 months after rectal surgery
  The QLQ-CR29 (Quality of life of rectal cancer patients with 29 questions) has five functional and 18 symptom scales. Scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms of the symptom scales.
Qualiy of life with EQ5D-5L | At 1, 6 and 12 months after rectal surgery
  Mean Score of the EQ-5D-5L Quality of Life The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).The questionnaire is a self-report survey that measures quality of life across 5 domains: : mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state
  - The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, numbered from 0 to 100.
  ( 100 means "the best health you can imagine" and 0 means "the worst health you
Digestive function with LARS score | At 1, 6 and 12 months after rectal surgery
  The LARS questionnaire (low anterior resection score) evaluates bowel function. Five questions regarding incontinence for flatus and liquid stools, frequency, clustering and urgency for defecation are taken into account. The score ranges from 0 to 42 is divides into no LARS (0 to 20 points), minor LARS (21 to 29 points), and major LARS (30 to 42 points).
Anal Incontinence with Wexner score ( or Vaizey score) | At 1,6 and 12 months after rectal surgery
  The WEXNER score assesses the importance of anal incontinence, it varies from 0 to 20, where 20 corresponding to total anal incontinence
  The Vaizey score assesses the importance of anal incontinence score from 0-28 where 0 means better outcomes
Female Sexual Function Index (FSFI) scale scores | At 1, 6 and 12 months after rectal surgery
  Measured in female patients. The Female Sexual Function Index (FSFI) is a 19-item self-report inventory designed to assess female sexual function. It comprises six domains: desire, arousal ,lubrication orgasm, satisfaction, pain. The maximum score for each domain is 6.0, obtained by summing item responses and multiplying by a correction factor. The total composite sexual function score is a sum of domain scores and ranges from 2.0 (not sexually active and no desire) to 36.0.
International Index of Erectile Function (IIEF)-5 | At 1,6 and 12 months after rectal surgery
  Measured in male patients
  IIEF assessment assesses to a limit the psychosexual background and the partner relationship, both considered important factors in the presentation of male sexual dysfunction.
  Scores of 0 to 5 are awarded to each of the 15 questions, then the scores are interpreted in the view of the5 domains from the original study.
  Domain A Erectile Function Domain B Orgasmic Function Domain C Sexual Desire Domain D Intercourse Satisfaction Domain E Overall Satisfaction
International Prostate Symptom Score (IPSS) | At 1, 6 and 12 months after surgery
  The International Prostate Symptom Score (I-PSS) is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life.
  Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom.
  The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
Predictive factors for anastomotic fistula | From the surgery to 12 months
  To identify predictive factors of anastomotic fistula from the surgery to 12 months
  Comparison of the clinical and perioperative data . The differences in proportions will be compared.

CONTACTS AND LOCATIONS:
Locations (15):
- Hôpital Universitaire de Belgique, Leuven, Belgium
- Canada (2):
  - Hôpital Universitaire McGill, Montreal
  - CHU de Quebec, Québec
- Hôpital Universitaire de Shanghai, Shanghai, China
- France (8):
  - CHU de Besançon, Besançon
  - Bordeaux Colorectal Institute, Bordeaux
  - Hôpital Bicêtre APHP, Le Kremlin-Bicêtre
  - CHU de Lyon, Lyon
  - Gp Hospitalier Diaconesses Croix St Simon, Paris
  - Hôpital Européen Georges Pompidou APHP, Paris
  - Hôpital Saint Antoine APHP, Paris
  - Hôpital Charles Nicolle, Rouen
- Policlinique Universitaire Gemelli, Roma, Italy
- Spain (2):
  - Hôpital General universitaire Madrid, Madrid
  - Hôpital Universitaire de Vigo, Vigo

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data(IPD) with other researchers.